CLINICAL TRIAL: NCT02083068
Title: Evaluation of the Protective Efficacy of a Vaccine Derived From the Synthetic CS Protein of Plasmodium Vivax
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Malaria Vaccine and Drug Development Center (Other)
Collaborators: The Administrative Department of Science, Technology and Innovation, Colciencias (Other)
Responsible Party: Principal Investigator, Socrates Herrera Valencia, MD, Malaria Vaccine and Drug Development Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2304-493-26202
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Malaria
Keywords: Malaria, vaccine, P. vivax
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): 10 individuals per sub- group to be immunized with the Vaccine PvCS N+C at month 0 and the Vaccine PvCS N+C+R at months 2 and 6
  Interventions: Biological: Vaccine PvCS N+C+R; Biological: Vaccine PvCS N+C
- Control (Placebo Comparator): six individuals for each sub- group to be immunized with placebo SSN Montanide ISA-51
  Interventions: Biological: SSN Montanide ISA-51

INTERVENTIONS:
Biological: Vaccine PvCS N+C+R — Vaccine PvCS N+C+R 60 mcg, freeze dried powder, Batch n°P0RGB, Exp: 18.10.2015 At month 2 and 6
  Arms: Experimental
Biological: Vaccine PvCS N+C — Vaccine PvCS N+C 60 mcg, freeze dried powder, Batch n°P0RGA, Exp: 18.10.2015, at month 0
  Arms: Experimental
Biological: SSN Montanide ISA-51 — SSN Montanide ISA-51 1 mL
  Arms: Control

SUMMARY:
This is a randomized, double-blind, controlled, which seeks to compare two groups of volunteers (naive and previously exposed to malaria) who were made 3 immunizations with a synthetic derivative of the CS protein of Plasmodium vivax in order to determine their protective efficacy. Then volunteers will be subject to an infectious challenge to assess the infectivity of gametocytes in the blood early stage of P. vivax in Anopheles albimanus mosquitoes.

DETAILED DESCRIPTION:
This study is a prospective controlled, blinded clinical trial, designed to establish the protective efficacy induced by the vaccine PvCSP between human volunteers with and without history of malaria.

Study subjects

This study will require the involvement of two types of volunteers:

* Parasite donors: 5-15 P. vivax-infected patients who will serve as parasites donors for experimental infection of mosquitoes, who will be enrolled in the endemic area.
* Volunteers for immunization: Two other groups of volunteers will be immunized with the vaccine PvCSP. A group of 16 people without previous exposure to malaria (naive) and another 16 people with a history of previous malaria infection (pre-immune).

Methodology Recruitment of infected patients: Parasite donors will be recruited among P. vivax infected patients attending a diagnostic center in the endemic area.

Infection of mosquitoes Blood from donors will be used to feed three days old mosquitoes by artificial membrane feeding technique. At day 7 a sample of mosquitoes will be examined to determine the degree of infection by dissection of the mosquito gut. On day 14, a small amount of mosquitoes with a good degree of infectivity will be used to infect challenged volunteers.

Recruitment of pre-immune and naive volunteers: Volunteers for the immunization stage will be recruited both in the city of Cali, non-endemic region, and in Buenaventura, a malaria endemic region, through various activities such as conferences, meetings and other means approved by the IRB like posters and flyers.

Immunization: Volunteers will be immunized with the vaccine (n=16) or placebo (n=16).

Follow Up Volunteers will be under medical vigilance during the first hour following the immunization to detect any adverse reaction. After the first hour period a medical exam will be made. Eight hours after immunization, each volunteer will be telephoned to assess physical condition. Any adverse event (AE) will be registered.

Subsequent follow up will be made on the day next to immunization and 1 or 2 weeks before the next immunization by a new clinical evaluation and AE report. Volunteers will be educated to contact the research staff at any moment.

Infection of volunteers Immunized volunteers will be challenged on day ~150 of the study, 1 month after the third immunization by the bite of 3±1 infected mosquitos. The "feeding cage" will be placed on the forearm of a volunteer for 10 minutes, allowing that the feeding window, wich will be covered by a mesh surface be placed against the volunteer's skin.

Volunteers will be educated about the signs and symptoms of malaria and they will have a daily telephone contact during the first 6 days.

Between days 7 and 23 the volunteers will be asked to go to the Clinical Trials Unit daily in order to establish the presence or absence of disease through thick blood smear and samples will be collected for retrospective real time PCR P. vivax.

From day 23 until day 31, volunteers will receive physical and laboratory evaluation every other day and will have daily telephone contact.

Once the patients present signs and symptoms of the disease curative treatment will be immediately provided, and 15 ml of blood will be drawn, which will be used for immune response assessment.

If the volunteers do not develop the disease during the follow-up period, on day 31 they will be given antimalarial treatment.

Treatment Volunteers will be treated with antimalarial drugs approved by the Colombian Ministry of Social Protection: chloroquine (three (3) doses: 600 mg initially, followed by 450mg at 24, and 48 hours), associated with primaquine (30mg/día) for 14 days. All the volunteers will be asked to return two weeks after starting treatment for a thick blood smear test to ensure cure of malaria.

ELIGIBILITY:
Inclusion Criteria:

* Naïve group

Healthy men and women aged 18-45 years. Signing freely and voluntary informed consent , accompanied by two witnesses who also sign.

Not have a history of malaria infection. For women, use of adequate contraception from the star restriction to be lifted by a doctor for contraception study. Accept not to travel to areas considered endemic for malaria during Trophies infectious period (1 month ) ( Buenaventura , Tierralta , Pretoria , Tumaco ,Urabá and Bajo Cauca) .

Be reachable by phone throughout the study period. Being Duffy positive ( Fy +) . Levels of hemoglobin ( Hb) > 11 g / dl. Availability to participate during the period in which they develop the study. Do not be participating in another clinical study

2. Preimmune group

Healthy men and women aged 18-45 years. Signing freely and voluntary informed consent , accompanied by two witnesses who also sign .

Having a history of infection (s ) and serological tests for malaria positive for P. vivax.

For women, use adequate contraception from the start restriction to be lifted by a doctor for contraception study .

Accept not to travel to areas considered endemic for malaria during Trophies infectious period (1 month ) ( Buenaventura , Tierralta , Pretoria , Tumaco Urabá and Bajo Cauca) .

Be reachable by phone throughout the study period. Availability to participate during the period in which they develop the study.

3. Voluntary blood donors

* Healthy men and women aged 18-45 years.
* Be positive diagnosis of P. vivax determined by thick smear examination .
* The patient must not have circulating malaria parasites such as P. falciparum or P. malariae .
* Have a parasitemia ≥ 0.1 %. by thick smear .
* Hb ≥ 9 g / dL at the time of diagnosis of malaria.
* The patient must have the capacity to provide informed consent freely and voluntarily . Should be illiterate may assert its decision to participate by putting their fingerprint in the format consent. Minors who are between 15 and 17 and wishing to participate must sign the informed consent and one of its Parents must sign the informed consent, accompanied by 2 witnesses who also sign

Exclusion Criteria:

* Step 1

  * Negative IFAT (< 1:20) for P. vivax on screening tests
  * Other criteria used in the case of naive volunteers, except a history of having lived in an endemic area for the past 6 months.

Step 2 Patients that have chronic or acute disease, different from malaria by P. vivax.

Having a history of disease or clinical conditions that according to medical criteria might increase significantly the risk related with participation on this study Hemoglobin levels <9 g/dL at the time of recruitment Have received antimalarial treatment before the diagnosis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Protective efficacy against P. vivax infection on volunteers exposed to infected mosquito bites | Thirty days after the last immunization
  Vaccine protective efficacy against P. vivax infection on volunteers exposed to infected mosquito bites

SECONDARY OUTCOMES:
Evolution of antibody titers | At months 0, 2, 4 and 6 of the trial
  Follow up every 2 months (month 0, 2, 4 and 6) until the end of the trial will be done to assess the evolution of P. vivax antibody titers.
Specific cytokine induction | At months 0, 2, 4 and 6 of the trial
  Specific cytokine induction will be measured by IFN- γ, TNF-α, IL-2; IL- 4, IL-6, IL-10
Changes on vaccine biological security | On the day next to immunization and 1 or 2 weeks before the next immunization
  Changes on vaccine biological security will be measured by renal, hepatic and hematologic function and pregnancy test.
Antibody functionality in vitro through inhibition of sporozoite invasion (ISI) to Hep-G2 cells. | Every 2 months
  Antibody functionality will be tested in vitro through essays of inhibition of sporozoite invasion (ISI) to Hep-G2 cells.
Vaccine-induced protection for P. vivax | 28 days after mosquito bites
  Vaccine-induced protection for P. vivax will be assessed by pre-patent period onset after infected mosquito bites exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Malaria Vaccine and Drug Development Center, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Background] Herrera S, Solarte Y, Jordan-Villegas A, Echavarria JF, Rocha L, Palacios R, Ramirez O, Velez JD, Epstein JE, Richie TL, Arevalo-Herrera M. Consistent safety and infectivity in sporozoite challenge model of Plasmodium vivax in malaria-naive human volunteers. Am J Trop Med Hyg. 2011 Feb;84(2 Suppl):4-11. doi: 10.4269/ajtmh.2011.09-0498. PMID 21292872
- [Derived] Arevalo-Herrera M, Gaitan X, Larmat-Delgado M, Caicedo MA, Herrera SM, Henao-Giraldo J, Castellanos A, Devaud JC, Pannatier A, Onate J, Corradin G, Herrera S. Randomized clinical trial to assess the protective efficacy of a Plasmodium vivax CS synthetic vaccine. Nat Commun. 2022 Mar 25;13(1):1603. doi: 10.1038/s41467-022-29226-3. PMID 35338131